CLINICAL TRIAL: NCT07353541
Title: An Evaluation of the Safety and Efficacy of a Standardized Diagnosis and Treatment Protocol for Esophageal Fistula in Patients With Esophageal Squamous Cell Carcinoma: A Single-Arm, Multi-Center Clinical Study
Brief Title: Standardized Management of Esophageal Fistula in Esophageal Squamous Cell Carcinoma
Acronym: PKU-ESCC-EF
Status: Not yet recruiting | Type: Observational
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Sponsor
Other Study IDs: PKU-ESCC-EF-ORS-001; 2024YJZ21 (Other: Peking University Cancer Hospital)
Record Dates: First submitted 2025-11-19; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-12

CONDITIONS: Esophageal Squamous Cell Carcinoma (ESCC); Esophageal Fistula
Keywords: Esophageal Squamous Cell Carcinoma; Esophageal Fistula; Standardized Management; Stent Placement; Nutritional Support; Observational Study; Registry Study; Real-world Evidence
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma; Esophageal Fistula

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples With DNA — Biospecimens to be retained include peripheral blood samples for complete blood count, biochemistry, coagulation function, thyroid function, and lymphocyte subset analysis, urine samples for routine urinalysis, and esophageal tissue specimens (two biopsies collected from the peri-fistula region during endoscopic procedures) for histopathological examination and biomarker profiling (EGFR, PD-L1, Ki67). All specimens will be collected, processed, and stored under standardized protocols by qualified investigators and clinical staff.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Standardized Management Cohort: All enrolled patients with advanced esophageal squamous cell carcinoma and newly diagnosed esophageal fistula who receive the standardized diagnosis and treatment protocol.
  Interventions: Other: Standardized Management Protocol for Esophageal Fistula

INTERVENTIONS:
Other: Standardized Management Protocol for Esophageal Fistula — This is a comprehensive, standardized clinical management protocol for esophageal fistula in advanced esophageal squamous cell carcinoma patients. The protocol integrates multiple standardized components into a unified pathway: (1) systematic diagnosis using iodine-contrast esophagography, chest CT, and endoscopy; (2) interventional fistula sealing with covered esophageal/airway stents selected by fistula characteristics; (3) coordinated adjunctive therapy including anti-infectives, acid suppression, and negative suction; (4) mandatory nutritional assessment with early transition from parenteral to enteral feeding; and (5) a defined pathway for subsequent anti-tumor therapy after clinical recovery. This multi-modal, sequential approach differentiates it from isolated interventions by providing integrated management from diagnosis through nutritional rehabilitation to subsequent oncology care within a standardized framework.

SUMMARY:
This prospective, multi-center, observational registry study (PKU-ESCC-EF) aims to evaluate the safety and effectiveness of a standardized diagnosis and treatment protocol for esophageal fistula (EF) in patients with advanced esophageal squamous cell carcinoma (ESCC). Esophageal fistula is a severe complication that often leads to life-threatening infections and poor nutrition. This study will observe patients receiving a comprehensive management strategy, which includes fistula sealing with esophageal or airway stents, targeted anti-infective therapy, nutritional support, and subsequent systemic anti-tumor therapy. The primary goal is to assess whether this standardized approach can improve overall survival and enable more patients to receive further anti-cancer treatments.

DETAILED DESCRIPTION:
This observational registry employs a prospective, single-arm design to recruit eligible patients with newly diagnosed esophageal fistula (tracheoesophageal or mediastinal fistula) complicating unresectable advanced esophageal squamous cell carcinoma. All enrolled participants will receive management according to a predefined standardized diagnostic and therapeutic protocol. The protocol integrates a comprehensive workflow from diagnostic assessment to multidisciplinary intervention: initial diagnosis is supported by clinical manifestations, imaging studies, and endoscopic evaluation, followed by interventional fistula closure using esophageal or airway covered stents selected according to fistula characteristics. Accompanying medical support includes anti-infective therapy, negative pressure suction, anti-reflux treatment, and nutritional support. After achieving adequate fistula control and clinical stabilization, subsequent systemic anti-tumor therapy may be administered based on investigator assessment. Prospective data collection will encompass fistula sealing status, nutritional parameters, quality of life, subsequent anti-tumor treatment rate, overall survival, and exploratory biomarker analysis of biospecimens, thereby providing real-world evidence to standardize management strategies for this serious complication.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary participation and provision of written informed consent.
* Age between 18 and 75 years (inclusive).
* Histologically confirmed diagnosis of esophageal squamous cell carcinoma.
* Radiologically confirmed unresectable, advanced disease.
* Newly diagnosed esophageal fistula (including tracheoesophageal fistula or mediastinal esophageal fistula).
* Previous receipt of ≤ 3 lines of systemic anti-tumor therapy.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.
* Adequate organ and marrow function within 7 days prior to potential anti-tumor treatment, as defined by:
* Hemoglobin ≥ 9.0 g/dL
* Absolute neutrophil count (ANC) ≥ 1.5 × 10⁹/L
* Platelet count ≥ 100 × 10⁹/L
* Total bilirubin (TBIL) ≤ 1.5 × the upper limit of normal (ULN)
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 × ULN (or ≤ 5 × ULN in the presence of liver metastases)
* Serum creatinine ≤ 1.5 × ULN
* Adequate cardiac, pulmonary, and renal function to be eligible for general anesthesia, with no contraindications to general anesthesia.

Exclusion Criteria:

* Patients with postoperative anastomotic fistula.
* Uncontrolled active bleeding.
* Presence of a concurrent primary malignancy other than esophageal carcinoma.
* Clinically significant cardiovascular disease, including but not limited to:
* Heart failure (NYHA Class III-IV)
* Uncontrolled coronary artery disease, cardiomyopathy, or arrhythmia
* Uncontrolled hypertension
* History of myocardial infarction within the past 1 year
* Neurological or psychiatric disorders that impair cognitive ability, including the presence of central nervous system metastases.
* Uncontrolled, active severe clinical infection ( > Grade 2 per NCI-CTCAE version 5.0) within 14 days prior to enrollment, including active tuberculosis (this is a contraindication for anti-tumor therapy, not for interventional procedures).
* Known or self-reported HIV infection, or active Hepatitis B or Hepatitis C.
* A history of interstitial lung disease (e.g., interstitial pneumonia, pulmonary fibrosis), or evidence of interstitial lung disease on baseline chest X-ray/CT.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of adult patients (aged 18-75 years) with unresectable, advanced esophageal squamous cell carcinoma (ESCC) who have been newly diagnosed with an esophageal fistula (tracheoesophageal or tracheomediastinal fistula). Eligible participants must have received no more than three prior lines of systemic anti-tumor therapy and must demonstrate adequate organ function and an Eastern Cooperative Oncology Group (ECOG) performance status of 0-2, making them potential candidates for subsequent anti-tumor treatment following fistula management. Patients with postoperative anastomotic leaks, other active malignancies, uncontrolled infections, significant cardiopulmonary disease, or other specified exclusion criteria will not be eligible for enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | From date of fistula diagnosis until death from any cause, assessed up to 6 months.
  Overall survival is defined as the time from the diagnosis of esophageal fistula to death from any cause

SECONDARY OUTCOMES:
Rate of Subsequent Anti-tumor Therapy | From date of fistula diagnosis until the initiation of subsequent anti-tumor therapy, assessed through study completion (up to 6 months).
  The proportion of patients who successfully receive/re-initiate systemic anti-tumor therapy after fistula control and clinical recovery.
Fistula Sealing Success Rate | At 2 weeks and 4 weeks after the initial fistula intervention.
  The success rate of fistula sealing, evaluated as either Complete Remission (CR) or Partial Remission (PR) according to the protocol's criteria.
Nutritional Status (NRS 2002) | From baseline through study completion (up to 6 months).
  Nutritional risk will be assessed using the Nutritional Risk Screening 2002 (NRS 2002) tool. The total NRS 2002 score is derived from the sum of three components:
  Nutritional Status Impairment Score (range: 0-3 points),
  Disease Severity Score (range: 0-3 points), and
  Age Adjustment (1 point if age ≥70 years; 0 points otherwise).
  The total score ranges from 0 to 7 points. A higher total score indicates a greater nutritional risk (i.e., a worse outcome). In accordance with the original validation, a total score of ≥3 points is considered indicative of nutritional risk.
Nutritional Status (PG-SGA) | From baseline through study completion (up to 6 months).
  Nutritional status will be assessed using the Patient-Generated Subjective Global Assessment (PG-SGA) tool. The PG-SGA yields two primary outcomes:
  1. Global Rating Categories: Patients are classified as Category A (Well nourished), Category B (Moderately malnourished or suspected of malnourishment), or Category C (Severely malnourished).
  2. Total PG-SGA Score: A quantitative score is calculated from patient-generated and professional assessment components. The total score ranges from 0 to approximately 35 points. A higher score indicates a worse nutritional status and outcome (i.e., greater risk or severity of malnutrition). In clinical practice, a score of 4 or higher typically triggers the need for nutritional intervention.
Quality of Life (QOL) | From baseline through study completion (up to 6 months).
  Quality of Life will be assessed using the Functional Assessment of Cancer Therapy - Esophageal Cancer subscale (FACT-E). The FACT-E is composed of the general cancer module (FACT-G) and an esophageal cancer-specific subscale. The total score ranges from 0 to 180 points. A higher score indicates a better quality of life (i.e., a better outcome).
Incidence of Adverse Events (AEs) | From the start of the standardized management protocol until 30 days after the last intervention or through study completion, whichever comes first.
  Safety and tolerability assessed by the incidence and severity of adverse events (AEs) and serious adverse events (SAEs), graded according to NCI CTCAE v5.0.

OTHER OUTCOMES:
Percentage of Participants with PD-L1 Positive Expression in Tumor Tissue | At baseline (time of fistula diagnosis).
  PD-L1 expression will be assessed in baseline tumor tissue samples via immunohistochemistry (IHC). The result will be reported as the percentage of tumor cells with positive membrane staining (e.g., using Tumor Proportion Score, TPS) and/or combined positive score (CPS), as appropriate.
EGFR Expression Level in Tumor Tissue | At baseline (time of fistula diagnosis).
  EGFR expression will be assessed in baseline tumor tissue samples via immunohistochemistry (IHC). The result will be reported using a standardized scoring system (e.g., H-score or percentage of positive cells).
Ki-67 Proliferation Index in Tumor Tissue | At baseline (time of fistula diagnosis).
  Ki-67 expression will be assessed in baseline tumor tissue samples via immunohistochemistry (IHC). The result will be reported as the Ki-67 proliferation index (percentage of positively stained tumor cell nuclei).

IPD SHARING:
Plan to Share IPD: Undecided